CLINICAL TRIAL: NCT03821623
Title: Nicotinamide Riboside Supplementation for Treating Elevated Systolic Blood Pressure and Arterial Stiffness in Middle-aged and Older Adults
Brief Title: Nicotinamide Riboside for Treating Elevated Systolic Blood Pressure and Arterial Stiffness in Middle-aged and Older Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Douglas Seals (Other)
Responsible Party: Sponsor-Investigator, Douglas Seals, Principal Investigator, University of Colorado, Boulder
Organization: University of Colorado, Boulder (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-0644
Record Dates: First submitted 2019-01-14; First posted 2019-01-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Aging
MeSH Terms: conditions — Hypertension | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotinamide riboside (Experimental): Subjects will take 500 mg of the vitamin B3-precursor, nicotinamide riboside (NIAGEN) twice per day (1,000 mg per day total) for 3 months.
  Interventions: Drug: Nicotinamide riboside
- Placebo (Placebo Comparator): Subjects will take placebo pills twice a day for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotinamide riboside — Nicotinamide riboside, a dietary supplement available over the counter under the name NIAGEN®, (ChromaDex Inc) is an exogenous NAD+ precursor that reverses age-related arterial dysfunction in aged mice, suggesting that declining NAD+ may play a key role in cardiovascular aging.
  Arms: Nicotinamide riboside
Other: Placebo — Subjects will take placebo pills twice a day for 3 months
  Arms: Placebo

SUMMARY:
Aging is the primary risk factor for cardiovascular diseases (CVD), the number one cause of death in developed societies. Systolic blood pressure (SBP) increase with age and is a key intermediary factor linking aging to increased CVD risk. The primary mechanisms underlying the age-associated increase in SBP is stiffening of the large elastic arteries, which is mediated by increases in oxidative stress, inflammation, and vascular smooth muscle tone. Regular caloric restriction is effective at lowering SBP in middle-aged and older adults; however, adherence to caloric restriction is poor and may be detrimental to normal weight older adults due to reduced skeletal muscle mass and bone mineral density. Therefore, identification of more practical alternative interventions that mimic the beneficial effects of caloric restriction, with stronger adherence and less risk of adverse consequences, is of significant biomedical importance.

Nicotinamide riboside is a naturally occurring precursor of nicotinamide adenine dinucleotide (NAD+), a critical mediator of the beneficial effects of caloric restriction, and therefore a novel caloric restriction mimetic compound. We recently completed the first pilot study of nicotinamide riboside supplementation in healthy middle-aged and older adults and demonstrated that 6 weeks of supplementation decreased systolic blood pressure (SBP) by 8 mmHg in individuals with baseline SBP of 120-139 mmHg (elevated SBP/stage 1 hypertension) compared with placebo, and lowered arterial stiffness, a strong independent predictor of CVD and related morbidity and mortality.

As a next translational step, we will conduct a randomized, placebo-controlled, double-blind clinical trial to further assess the safety and efficacy of oral nicotinamide riboside (3 months vs placebo) for decreasing SBP and arterial stiffness in middle-aged and older men and women with SBP between 120 and 139 mmHg at baseline.

DETAILED DESCRIPTION:
Study Overview: This is a randomized, double-blind, placebo-controlled, parallel design, single site phase IIa clinical trial assessing the efficacy of nicotinamide riboside supplementation to lower systolic blood pressure (SBP) and aortic stiffness in middle-aged to older (MA/O) adults (50-79 years) with elevated to stage-1 systolic hypertension (SBP: 120-139 mmHg). Nicotinamide riboside is an endogenously occurring precursor of NAD+ and a novel caloric restriction mimetic in humans that is now commercially available as a dietary ingredient/supplement. We have recently demonstrated that chronic supplementation with nicotinamide riboside lowers SBP and carotid-femoral pulse wave velocity (CFPWV; gold-standard measure of aortic stiffness and independent risk factor for cardiovascular diseases) in a small pilot study of healthy MA/O adults; the greatest reductions in SBP were observed in a subgroup with baseline SBP in the elevated/stage-1 hypertension range. As a next translational step, the present study proposes to assess the efficacy of 3 months of nicotinamide riboside supplementation for decreasing SBP (primary outcome) and aortic stiffness (secondary outcome) in a larger cohort of MA/O men and women with SBP in the elevated/stage-1 hypertension range. As secondary aims, we will also assess safety and tolerability of long-term nicotinamide riboside supplementation, and the effects of nicotinamide riboside supplementation vs. placebo on NAD+ metabolites and circulating biomarkers of vasoconstriction, oxidative stress and inflammation.

Subject Enrollment and Screening: Potential participants will be made aware of the proposed study through described recruitment efforts (see Recruitment and Retention section). Interested participants will contact a staff research assistant via phone or email (contact information supplied with recruitment materials) and will complete a general screening form online through the Research Electronic Data Capture (REDCap) system to determine eligibility. REDCap is a secure web-based application designed to support data capture for research studies.

After hearing a thorough study description and having all questions answered by the staff research assistant, those eligible and interested in participating in the study will provide written and verbal informed consent, and undergo in-person screening at the CU Boulder Clinical Translational Research Center (CTRC). Informed consent will only be obtained by members of the research team who have been observed and approved by the CTRC Research Subject Advocate (see Protection of Human Subjects). We plan to consent 148 subjects in order to meet our enrollment targets (to account for an ~25% rate of exclusion base on in-person screening).

In-person screening will include: review of medical history; physical exam; resting heart rate; resting blood pressure; blood draw for metabolic profile, lipid profile, complete blood count, and thyroid stimulating hormone; measurement of ankle-brachial index; and a 12-lead ECG at rest and during graded exercise testing (see the Eligibility Criteria section for detailed inclusion/exclusion criteria).

Resting blood pressure will be measured on a second occasion within one week of the initial screening to establish baseline blood pressure status; SBP measured on the two separate days will be averaged and must be in the elevated to stage-1 hypertension range (120-139 mmHg) for enrollment into the study.

Participant Randomization and Subject/Investigator Blinding: After completing screening, eligible subjects will be randomized to either the nicotinamide riboside or placebo group. A randomized block design will be used to balance groups for sex, age (mid-life: 50-64 years vs. older: 65-79 years) and hypertension status (elevated vs. stage-1 systolic hypertension). Randomization will be carried out by an unblinded staff research assistant who is not involved in data collection or analysis. Subjects will be categorized based on the block randomization scheme and then a random number generator will be used to assign subjects to either nicotinamide riboside or placebo treatment. Researchers involved in collection of outcome data will be blinded to the assigned intervention. Subjects will be blinded to their assigned intervention and will receive capsules in coded blister packs; nicotinamide riboside and placebo capsules will appear identical. CTRC clinical staff involved with subject check-in visits and/or data collection will also be blinded (in the case of a serious adverse event, blinding of the CTRC staff will be broken, as necessary to ensure appropriate medical treatment).

Assessment of Study Outcomes: All subjects will undergo baseline testing for all primary, secondary, and other outcome measures. All measurements will be made after a 12 hour fast from food and caffeine (water allowed) and 24 hours after abstaining from alcohol and exercise. All tests will take place in the CU Boulder CTRC.

The protocol for baseline testing is as follows:

* Urine sample collection;
* Assessment of casual SBP;
* Placement of IV in an antecubital vein followed by 30 minutes of rest in a supine position; - Collection of blood samples by a trained CTRC provider;
* Assessment of aortic stiffness by CFPWV.

Following completion of outcome measure testing, the below non-outcome measures will be made in order to ensure that participant characteristics known to affect cardiovascular function are unaltered during the intervention:

* 3-day diet records to ensure that daily fluid and caloric intake remain stable;
* The Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire will be completed and physical activity will be assessed by accelerometers (ActiGraph, 3-day recordings) to document stability of physical activity levels;
* Maximal oxygen consumption using indirect calorimetry during incremental treadmill exercise (Balke protocol) will be measured to document unchanged aerobic fitness; and
* Body composition will be assessed by dual energy x-ray absorptiometry (DEXA) and anthropometry to confirm unaltered body composition; body mass will also be determined during safety and check in visits with CTRC nursing staff.

Following all CTRC testing procedures, subjects will be outfitted with an ambulatory blood pressure monitor pre-programmed to automatically measure blood pressure every 20 minutes. A study team member will provide the subject with written and verbal instructions on how to operate the monitor. Subjects will wear the monitor for 24 hours before returning it to the investigators. Ambulatory blood pressure data will be evaluated for completeness immediately upon return of the monitor; if an inadequate number of blood pressure measurements (<67% of expected) were made to properly characterize 24-hour SBP the subject will be re-outfitted with the ambulatory monitor, be re-instructed on its use, and wear it for a second 24-hour period.

The Research Strategy and Outcome Measures sections provide a more detailed description of these procedures. Similar protocols and procedures are well established in the Seals laboratory and the CU Boulder CTRC.

Delivery of the Intervention: After completing baseline testing, subjects will begin their assigned intervention (nicotinamide riboside or placebo). Subjects will be instructed to take 2 x 250 mg capsules in the morning and 2 x 250 mg capsules in the evening (4 capsules/day). This will result in a dosing of 500 mg nicotinamide riboside 2x/day in the nicotinamide riboside group (1000 mg/day total).

Subjects will return to the CU Boulder CTRC once every two weeks for check-in and to receive capsules. Capsules will be prepared by the manufacturer in blister packs to promote adherence and will be stored and dispensed by the CTRC pharmacist (unblinded) and distributed by a CTRC nurse (blinded). Subjects will return their blister packs at each check-in visit and after follow-up testing to assess adherence to the intervention. During each visit to the CTRC, subjects will be monitored for treatment-emergent adverse events by blinded CTRC clinical staff.

Post-Testing: After completing 3 months of treatment with either nicotinamide riboside or placebo, subjects will return to the CU Boulder CTRC for reassessment of all outcome measures, including: casual SBP, 24-h ambulatory SBP, CFPWV, venous blood draw, and urine sample. Non-outcome control measures (3-day diet record, CHAMPS survey, activity monitor, maximal oxygen consumption test, body composition) will also be reassessed. These measures will be made under the same experimental conditions, in the same order, and with the same techniques as baseline testing.

Intervention Duration and Study Sample Size: The expected duration for a participant to complete the entire protocol from screening to follow-up testing is 18 weeks. Based on our power analysis, we need to complete the entire protocol on a total of 94 participants (47/group) to detect a significant difference between treatment conditions in our primary outcome measure (SBP). We intend to enroll 118 subjects (59/group) to account for an ~20% dropout rate. Based on this, we will enroll 2-3 subjects per month, which will allow for completion of data collection by month 55 of this award; this rate of testing is achievable based on previous pharmacological interventions carried out in the Seals laboratory and the availability of the CTRC facilities and staff.

Data Collection and Analysis (including blinding): Collection of primary and secondary outcome measures will be performed by postdoctoral fellow, Dr. Craighead, with the assistance of members of the laboratory. IV placement and blood draws will be performed by experienced CTRC clinical staff. Data analysis will be performed by Dr. Craighead. Having a single investigator perform all data collection and analysis will remove the potential for inter-investigator variation. Dr. Craighead and other research and clinical staff involved in data acquisition will remain blinded throughout data collection and analysis. All data will be analyzed as outlined in the Research Strategy section and Outcome Measures section; data analysis and dissemination of results will be completed by the end of this award.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Willing to accept random assignment to condition
* Systolic blood pressure between 120 and 159 mmHg
* Body mass index <40 kg/m2
* Weight stable in the prior 3 months (<2 kg weight change) and willing to remain weight stable throughout the study
* Absence of other clinical disease as determined by medical history, physical examination, blood chemistries, ankle-brachial index, and 12-lead ECG at rest and during graded treadmill exercise

  * Ankle-brachial index >0.7
  * Total cholesterol <240 mg/dL
  * Fasting plasma glucose <126 mg/dL
  * Normal 12-lead ECG at rest and during graded treadmill exercise to fatigue

Exclusion Criteria:

* Systolic blood pressure <120 or >/= 160 mmHg
* Currently taking antihypertensive medications
* Other chronic medical condition (e.g., diabetes, chronic kidney disease, cancer)
* Current smoker
* Alcohol dependence or abuse
* Uncontrolled thyroid disease or change in thyroid medication within previous 3 months
* Abnormal blood pressure response to exercise (drop in SBP below resting pressure or SBP >160 mmHg or DBP >115 mmHg)
* Regular vigorous aerobic/endurance exercise (>4 bouts/weeks, >30 min/bout at a workload >6 METS)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 months
  Resting systolic blood pressure

SECONDARY OUTCOMES:
Ambulatory blood pressure | 3 months
  24-hour mean blood pressure
Arterial stiffness | 3 months
  Carotid-femoral pulse wave velocity

OTHER OUTCOMES:
Number and severity of adverse events (safety) | 3 months
  Monitoring and documentation of number and type of adverse events
Number of participants that dropout due to adverse events (tolerability) | 3 months
  Monitoring subject dropout due to adverse events
Adherence to the intervention (percentage of prescribed pills consumed) | 3 months
  Counting returned pills on a bi-weekly basis to determine what percentage of prescribed pills subjects take.
NAD+ and related metabolite blood levels | 3 months
  Blood samples will be analysed using high performance liquid chromatography-mass spectronomy analysis for levels of NAD+ and related metabolites including: NADP+, nicotinic acid adeniene dinucleotide, nicotinamide, and nicotinamide mononucleotide.
Sympathetic activity | 3 months
  Plasma norepinephrine, a marker of sympathetic activity, will be measured by high performance liquid chromatography
Oxidative stress | 3 months
  Plasma oxidized LDL, a marker of oxidative stress, will be measured by ELISA
Inflammation | 3 months
  Plasma interleukin-6, a marker of inflammation, will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Physiology of Aging Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martens CR, Denman BA, Mazzo MR, Armstrong ML, Reisdorph N, McQueen MB, Chonchol M, Seals DR. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun. 2018 Mar 29;9(1):1286. doi: 10.1038/s41467-018-03421-7. PMID 29599478
- [Derived] Oh ES, Opoku G, Darvish S, Craighead DH, Ostrow A, Rossman MJ, Steele CN, Struemph T, You Z, Seals DR, Chonchol M, Nowak KL. Sex Differences in Dementia and Mild Cognitive Impairment in Nondialysis CKD. Clin J Am Soc Nephrol. 2025 Nov 20. doi: 10.2215/CJN.0000000922. Online ahead of print. No abstract available. PMID 41264372
- [Derived] Freeberg KA, Craighead DH, Martens CR, You Z, Chonchol M, Seals DR. Nicotinamide Riboside Supplementation for Treating Elevated Systolic Blood Pressure and Arterial Stiffness in Midlife and Older Adults. Front Cardiovasc Med. 2022 May 10;9:881703. doi: 10.3389/fcvm.2022.881703. eCollection 2022. PMID 35620522